CLINICAL TRIAL: NCT03690947
Title: Randomized, Double-blinded, Controlled Clinical Trial of Combination of Intravitreal Ranibizumab With or Without Micropulse Laser for the Treatment of Diabetic Macular Edema
Brief Title: Combination of Intravitreal Ranibizumab With or Without Micropulse Laser for the Treatment of DME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Yu Xiaobing, M.D., Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z181100001718079
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy Group (Experimental)
  Interventions: Drug: Intravitreal Ranibizumab; Procedure: Micropulse Laser
- Intravitreal Ranibizumab Group (Active Comparator)
  Interventions: Drug: Intravitreal Ranibizumab; Drug: Intravitreal Ranibizumab as needed

INTERVENTIONS:
Drug: Intravitreal Ranibizumab — All subjections received 3 initial Ranibizumab injections
  Other Names: Lucentis
Procedure: Micropulse Laser — After 3 initial Ranibizumab injections, Micropulse Laser will be done as needed each month if macular edema persists
  Other Names: Macular Laser Photocoagulation
  Arms: Combination Therapy Group
Drug: Intravitreal Ranibizumab as needed — After 3 initial Ranibizumab injections, Ranibizumab will be injected as needed till BCVA reaches stabilization
  Other Names: Lucentis
  Arms: Intravitreal Ranibizumab Group

SUMMARY:
The objective of this study is to evaluate if combination of intravitreal ranibizumab with micropulse laser shows non inferiority compared to intravitreal ranibizumab only in diabetic macular edema.

DETAILED DESCRIPTION:
To investigate the efficacy of intravitreal ranibizumab injections compared to combination with Micropulse Laser in Chinese patients with visual impairment in DME.

The result of the study will be used to support new therapy in DME patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form must be signed before any tests or procedures are done
* Male or female of 30 to 80 years of age (inclusive) at the first screening visit
* Diagnosis of type 2 diabetes, with fasting blood glucose≤10mmol/L, HbA1C≤10.0%
* Diabetic medication must be stable for at least 3 months before first screening visit and remain stable during study
* Diagnosis of non-proliferative diabetic retinopathy with diabetic macular edema resulting in visual acuity reduction
* Study eye's BCVA between 24 to 78 ETDRS letters at screening and baseline of the study
* Macular edema of the study eye and central retinal thickness ≥300 µm determined by SD-OCT
* Study eye had not had grid pattern photocoagulation, intraocular surgery, intravitreal corticosteroid injections and intravitreal anti-VEGF injections for at least 3 months before baseline
* Non-study eye's BCVA ≥ 24 ETDRS letters at screening and baseline of the study
* Non-study eye had not had intravitreal anti-VEGF injections for at least 3 months before baseline
* If both eyes qualify, then investigators will choose an eye with worse BCVA as study eye. Only study eye will receive intravitreal ranibizumab and/or Micropulse Laser treatment

Exclusion Criteria:

* Failure to follow study or follow-up procedures
* Pregnant or breast-feeding woman and woman without adequate method of contraception
* History of stroke or myocardial infarction within 3 months before screening
* Renal failure or creatinine > 2.0 mg/dl
* Uncontrolled systemic diseases or systemic treatment that may affect results of the study
* Active ocular or intraocular infections of either eye
* Neovascularization of the iris or neovascular glaucoma of either eye
* A history of uveitis or vitreous macular traction in study eye
* Glaucoma or IOP≥24 mmHg of study eye

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity changes | 12 months
  Compare the changes of BCVA between two groups

SECONDARY OUTCOMES:
Central Macular Thickness changes | 12 months
  Compare the changes of CMT between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Yu, M.D., Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Email yuxiaobing@sina.com for individual participant data
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Mi X, Gu X, Yu X. The efficacy of micropulse laser combined with ranibizumab in diabetic macular edema treatment: study protocol for a randomized controlled trial. Trials. 2022 Sep 2;23(1):736. doi: 10.1186/s13063-022-06593-2. PMID 36056443